CLINICAL TRIAL: NCT05146869
Title: A Randomized, Open-Label, Parallel-Cohort, Single-dose and Multiple-dose Phase I Study of DBPR108 Tablets in Type 2 Diabetes Mellitus Patients
Brief Title: A Single-dose and Multiple-dose Study to Evaluate the Pharmacokinetics and Pharmacodynamics of DBPR108 Tablets in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA1118-014
Record Dates: First submitted 2021-11-12; First posted 2021-12-07 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — DBPR108

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 50 mg DBPR108 tablets (Experimental): 10 patients will be randomized to receive 50 mg DBPR108 tablets.
  Interventions: Drug: DBPR108 tablets
- 100 mg DBPR108 tablets (Experimental): 10 patients will be randomized to receive 100 mg DBPR108 tablets.
  Interventions: Drug: DBPR108 tablets
- 200 mg DBPR108 tablets (Experimental): 10 patients will be randomized to receive 200 mg DBPR108 tablets.
  Interventions: Drug: DBPR108 tablets

INTERVENTIONS:
Drug: DBPR108 tablets — DBPR108 tablets, oral, once daily on Day 1 and Day 3-9 for a total of 8 doses.

SUMMARY:
This is a phase I study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single-dose and multiple-dose of DBPR108 tablets in Type 2 Diabetes Mellitus Patients.

DETAILED DESCRIPTION:
This study aims to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics characteristics, single-dose and multiple-dose of DBPR108 tablets in Chinese Type 2 Diabetes Mellitus Patients. The 30 eligible patients will be randomized to receive 50 mg, 100 mg, or 200 mg DBPR108 tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the World Health Organization (WHO) (1999) criteria for the diagnosis and classification criteria for type 2 diabetes mellitus;
2. 18 ≤ age ≤ 75 years old, male or female;
3. Body mass index (BMI) within the range of 19-35 kg/m^2 (inclusive), BMI = weight (kg) / height^2 (m^2);
4. 7.0% ≤Hemoglobin A1c (HbA1c) ≤ 9.5%;
5. Patients who voluntarily participate in the study and sign the informed consent form;
6. Patients who agree to use contraception from the signing of the informed consent form until 1 month after the end of the last medication.

Exclusion Criteria:

1. Fasting plasma glucose (FPG) > 13.9 mmol/L;
2. The investigator determines that the patients need to use insulin therapy;
3. Patients with acute or serious complications of diabetes (including diabetic ketoacidosis, hyperosmotic nonketotic diabetic coma, lactic acidosis and hypoglycemia coma);
4. History of severe hypoglycemia (hypoglycemia with severe cognitive impairment and requiring other measures to help recover);
5. History of acute or chronic pancreatitis, or related diseases that are most common cause of acute pancreatitis (such as recurrent cholelithiasis, etc.);
6. History of allergy to DPP-4 inhibitors or the investigator determines that the patients may be allergic to investigational drug;
7. Patients with untreated hyperthyroidism and other diseases, which may affect blood glucose;
8. Patients who have used other hypoglycemic drugs within 14 days before the first dose; or patients who are not suitable for this study as determined by the investigator due to taking other hypoglycemic drugs;
9. Patients with inflammatory bowel disease, partial intestinal obstruction or chronic bowel disease related to obvious digestive and absorption disorders;
10. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 3 * upper limit of normal (ULN), or total bilirubin > 1.5 *ULN;
11. Abnormal renal function: serum creatinine>1.5 * ULN; or eGFR< 45 mL/min/1.73m^2;
12. White blood cells (WBC) < 3.0 *10^9/L and neutrophil count of peripheral blood < 1.5 * 10^9/L; hemoglobin < 100 g / L; triglyceride > 5.7 mmol/L;
13. Patients who have the second or third degree atrioventricular block, long Q-T syndrome, or QTc>500 ms without cardiac pacemaker;
14. Patients with any one of HBsAg, hepatitis C antibody, anti-HIV antibody and antibody of treponema pallidum positive;
15. Female patients of childbearing age with pregnant test positive or lactating women;
16. History of alcohol or drug abuse within 3 months before screening, alcohol abuse is average alcohol intake more than 14 units alcohol (1 unit=12 ounces or 360 mL of beer,1.5 ounces or 45 mL spirits with 40% alc/vol, 5 ounces or 150 mL grape wine); or intake any other products containing alcohol within 2 days before the first administration of investigational product;
17. Patients who smoke more than 5 cigarettes per day within 3 months prior to screening;
18. Patients with consumption of grapefruit juice, methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks) within 2 days before the first administration in treatment period , or patients who have strenuous exercise, or have other factors affecting drug absorption, distribution, metabolism, excretion, etc;
19. Participation in other clinical trials or administration of any other investigational drugs or devices within 3 months before screening;
20. Patients with the following diseases:

    1. Serious dysrhythmias, obvious left ventricular dysfunction, New York Heart Association (NYHA) functional class III or IV;
    2. History of unstable angina pectoris, myocardial infarction, or other high-risk coronary artery diseases;
    3. Uncontrolled hypertension, systolic pressure ≥160 mmHg or diastolic pressure ≥100 mmHg;
    4. History of cancer , organ transplantation;
    5. History of epilepsy, psychosis, severe depression, etc.
21. Not suitable for this study as determined by the investigator due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of DBPR108 tablets | Day 1-Day 11
  Cmax of DBPR108 tablets will be assessed after single-dose and multiple-dose administration
Area under the plasma concentration versus time curve (AUC) of DBPR108 tablets in plasma | Day 1-Day 11
  AUC of DBPR108 tablets will be assessed after single-dose and multiple-dose administration
Half-life(t1/2) of DBPR108 tablets | Day 1-Day 11
  T1/2 of DBPR108 tablets will be assessed after single-dose and multiple-dose administration
Apparent volume of Distribution(Vz/F)of DBPR108 tablets | Day 1-Day 11
  Vz/F of DBPR108 tablets will be assessed after single-dose and multiple-dose administration
CL/F of DBPR108 tablets | Day 1-Day 11
  Apparent clearance(CL/F) of DBPR108 tablets will be assessed single-dose and multiple-dose administration
Change from baseline in dipeptidyl peptidase-IV inhibition rate | Day 1-Day 11
  Change from baseline in dipeptidyl peptidase-IV inhibition rate will be assessed after single-dose and multiple-dose administration
Change from baseline in active glucagon-like peptide1 concentration | Day 1-Day 11
  Change from baseline in active glucagon-like peptide1 concentration will be assessed after single-dose and multiple-dose administration

SECONDARY OUTCOMES:
The number of patients with adverse events | Throughout the study period, with an average of 1 months
  The number of patients with adverse events as a measure of safety and tolerability.
Clinically significant changes from baseline in 12-lead electrocardiogram (ECG) examination will be recorded as AEs at each visit time point | Within screening period (Day-21 to Day-15), baseline period (Day-7 to Day-1), and before discharge (Day11).
  ECG monitoring includes P-R, QT and QTc intervals in ms.
Clinically significant changes from baseline in vital signs examination will be recorded as AEs at each visit time point. | Throughout the study period, with an average of 1 months
  Vital signs monitoring includes respiratory rate and pulse in times per minute
Clinically significant changes from baseline in vital signs examination will be recorded as AEs at each visit time point. | Throughout the study period, with an average of 1 months
  Vital signs monitoring includes systolic blood pressure and diastolic blood pressure in mmHg.
Clinically significant changes from baseline in vital signs examination will be recorded as AEs at each visit time point. | Throughout the study period, with an average of 1 months
  Vital signs monitoring includes body temperature in degrees Celsius
Clinically significant changes from baseline in physical examination will be recorded as AEs at each visit time point. | Within screening period (Day-21 to Day-15), baseline period (Day-7 to Day-1), and before discharge (Day11).
  Physical examination includes mucocutaneous, lymphonodus, head and neck,chest, abdomen, spinal column, musculoskeletal, nervous system
Clinically significant changes from baseline in routine blood test will be recorded as AEs at each visit time point. | Within screening period (Day-21 to Day-15), baseline period (Day-7 to Day-1), and before discharge (Day11)
  Routine blood test includes white blood cell count, platelet, neutrophilic granulocyte count, lymphocyte count and monocyte count in 10^9 /L.
Clinically significant changes from baseline in blood biochemistry test will be recorded as AEs at each visit time point.recorded as AEs at each visit time point. | Within screening period (Day-21 to Day-15), baseline period (Day-7 to Day-1), and before discharge (Day11)
  Blood biochemistry test includes total protein, albumin and albumin in g/L.
Clinically significant changes from baseline in blood biochemistry test will be recorded as AEs at each visit time point.recorded as AEs at each visit time point. | Within screening period (Day-21 to Day-15), baseline period (Day-7 to Day-1), and before discharge (Day11)
  Blood biochemistry test includes alanine aminotransferase, aspartate aminotransferase, amylase, alkaline phosphatase and in U/L.
Clinically significant changes from baseline in blood biochemistry test will be recorded as AEs at each visit time point.recorded as AEs at each visit time point. | Within screening period (Day-21 to Day-15), baseline period (Day-7 to Day-1), and before discharge (Day11)
  Blood biochemistry test includes ureophil, glucose, triglyceridein, total cholesterol, high-density lipoprotein, low-density lipoprotein, sodium, potassium, chlorine, calcium in mmol/L
Clinically significant changes from baseline in blood biochemistry test will be recorded as AEs at each visit time point.recorded as AEs at each visit time point. | Within screening period (Day-21 to Day-15), baseline period (Day-7 to Day-1), and before discharge (Day 11)
  Blood biochemistry test includes total bilirubin and serum creatinine in umol/L.
Clinically significant changes from baseline in routine urine test will be recorded as AEs at each visit time point. | Within screening period (Day-21 to Day-15), baseline period (Day-7 to Day-1), and before discharge (Day11)
  Routine urine test includes the count of leukocyte, and red blood cell in high-power field.
Clinically significant changes from baseline in routine urine test will be recorded as AEs at each visit time point. | Within screening period (Day-21 to Day-15), baseline period (Day-7 to Day-1), and before discharge (Day11)
  Routine urine test includes glucose, protein, ketonein in negative or positive.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lin, PhD, Principal Investigator — Beijing Anzhen Hospital of Capital Medical University , Beijing, China; Shan NA Jing, PhD, Principal Investigator — Beijing Anzhen Hospital of Capital Medical University , Beijing, China
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu W, Yang K, Lin Y, Lu C, Liu J, Zhou H, Wang J, Zhang T, Yao L, Qi H, Zhang X, Jia R, Li X, Jing S. Pharmacokinetics and Pharmacodynamics of Prusogliptin (DBPR108), a Once-Daily Dipeptidyl Peptidase-4 Inhibitor, in Patients with Type 2 Diabetes. Clin Pharmacokinet. 2025 May;64(5):703-713. doi: 10.1007/s40262-025-01501-8. Epub 2025 Apr 19. PMID 40252162